CLINICAL TRIAL: NCT02816424
Title: Prevention of Teen Pregnancy Through Screening and Brief Intervention in Primary Care
Brief Title: Brief Intervention for Teen Pregnancy Prevention
Acronym: TEMPO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Collaborators: Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: TP2AH000028
Record Dates: First submitted 2016-06-09; First posted 2016-06-28 (Estimated); Last update posted 2022-05-24 (Actual); Status verified 2020-04

CONDITIONS: Teen Pregnancy Prevention
Keywords: Screening and Brief Intervention; Motivational Interviewing; Teen Pregnancy Prevention

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Brief Motivational Interviewing (Experimental): Principles and skills of motivational interviewing will be used with participants assigned to brief intervention. These participants will receive feedback that they are at risk for unintended pregnancy. They will receive information on the likelihood of pregnancy given their self-reported frequency of unprotected sex. They will be given information regarding negative consequences associated with teen pregnancy. They will be provided with information on the chances of pregnancy with abstinence, condom use, oral contraceptives, and Long Acting Reversible Contraceptives (LARC). Following information exchange, participants who are high in readiness to change will engage in action planning, whereby a specific plan for reducing risk for unintended pregnancy will be collaboratively developed with the interventionist. Patients who are low in readiness to change will complete a motivational interviewing-based roadmap activity that is designed to strategically evoke motivational speech.
  Interventions: Behavioral: Teens Exploring and Managing Prevention Options (TEMPO)
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Teens Exploring and Managing Prevention Options (TEMPO)
  Arms: Brief Motivational Interviewing

SUMMARY:
Although the Academy of Pediatrics and the Society for Adolescent Health and Medicine recommend that teen health providers screen for sexual risk behaviors and provide education and counseling to those at risk, there are currently no specific guidelines or protocols available to guide such practices, nor have there been any rigorous evaluations of efficacy. Preventing teen pregnancy through brief intervention in primary care holds the promise to have a significant public health impact and reduce health disparities by engaging, educating, and motivating the majority of teens who visit a primary care setting each year. In the current study, we seek to rigorously evaluate the impact of brief intervention vs. informational control on unprotected sexual intercourse among teens with past year unprotected sex at two primary care clinics serving predominately underserved, minority populations in New Mexico. The target population for the current study will be 1350 male and female teens, aged 13-19, from the Atrisco Center for Family and Community Health and the Albuquerque Job Corps Wellness Center. Extensive formative work involving the study population will be conducted prior to the trial to refine the motivational interviewing-based brief intervention. Eligible youth will be randomly assigned to brief intervention or an informational control condition, in addition to regularly offered medically-based contraception consultation and prescription services. Follow-ups at 3- and 9- months will compare rates of unprotected sex and acceptance of long-acting reversible contraceptives. Brief education and counseling interventions could be feasibly implemented during the greater than eight preventive and acute primary care visits that the average US adolescent attends during their teen years. Such an approach could conserve valuable resources required by more intensive interventions for nonresponsive teens with greater need. Furthermore, social determinants of health, such as poverty and race, that may reduce access to more extensive psychosocial interventions, are less likely to prevent access to primary care, increasing health equity.

ELIGIBILITY:
Inclusion Criteria:

* Aged 13-19
* Self-reported past year unprotected sex
* Can read and speak English
* Willing to be contacted for follow-up

Exclusion Criteria:

* Current use of long-acting reversible contraceptives
* Self-reported pregnancy or pregnancy discovered during optional medical contraception consultation
* Expressed suicidality
* Obvious cognitive impairment
* Inability to provide informed consent

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 447 (Actual)
Dates: Start 2015-11-11 (Actual); Primary Completion 2021-08-20 (Actual); Study Completion 2021-08-20 (Actual)

PRIMARY OUTCOMES:
Proportion of participants endorsing unprotected sex at 3 month follow up | 3-Month Endpoint
  All participants
Proportion of participants endorsing acceptance of Long Acting Reversible Contraception (LARC) at 3 month follow up | 3-Month Endpoint
  Among female participants

SECONDARY OUTCOMES:
Proportion of participants endorsing unprotected sex at 9 month follow up | 9-Month Endpoint
  All participants
Proportion of participants endorsing acceptance of Long Acting Reversible Contraception (LARC) at 9 month follow up | 9-Month Endpoint
  Among female participants

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer E Hettema, PhD, Principal Investigator — The University of New Mexico
Locations (1):
- The University of New Mexico, Albuquerque, New Mexico, United States